CLINICAL TRIAL: NCT05249101
Title: A Phase 1b/2, Dose-escalation, Randomized, Multicenter Study of Maintenance Ivaltinostat Plus Capecitabine or Capecitabine in Patients With Metastatic Pancreatic Adenocarcinoma Whose Disease Has Not Progressed on FOLFIRINOX
Brief Title: A Study of Ivaltinostat Plus Capecitabine or Capecitabine in Metastatic Pancreatic Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CG Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CG-745-2-08
Record Dates: First submitted 2022-01-29; First posted 2022-02-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — N1-(3-(dimethylamino)propyl)-N8-hydroxy-2-((naphthalene-1-loxy)methyl)oct-2-enediamide; Capecitabine

STUDY DESIGN:
Intervention Model Description: In Phase 1b, 3 dose levels of ivaltinostat will be studied in combination with a fixed dose of capecitabine to determine the RP2D of ivaltinostat.
  In Phase 2, patients will be randomized in a 1:1 ratio to the combination of ivaltinostat and capecitabine or to capecitabine monotherapy. A fixed dose for capecitabine 1000 mg/m2 orally twice daily will be taken on Days 1 to 14, and the RP2D of ivaltinostat will be administered intravenously once a week for 2 weeks, followed by 1 week of rest. One cycle consists of 21 days. Tumor response during study treatment will be assessed every 6 weeks up to Cycle 10, then every 9 weeks afterwards using RECIST v1.1 criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ivaltinostat plus Capecitabine (Experimental): Ivaltinostat plus Capecitabine
  Interventions: Drug: Ivaltinostat; Drug: Capecitabine
- Capecitabine Monotherapy (Active Comparator): Capecitabine Monotherapy
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Ivaltinostat — Ivaltinostat (E)-N1-(3-(dimethylamino)propyl)-N8-hydroxy-2-((naphthalen-1-yloxy)methyl)oct-2-enediamide phosphate) is a novel anticancer therapeutic candidate that inhibits enzymatic activity of histone deacetylase (HDAC).
  Arms: Ivaltinostat plus Capecitabine
Drug: Capecitabine — Capecitabine is labeled for monotherapy for the treatment of adjuvant Dukes' C colon cancer and metastatic colon cancer at a recommended dose of 1250 mg/m2 twice daily for 2 weeks followed by a 1-week rest. This dose schedule was effective and tolerable in the first line setting for patients with pancreatic cancer (Cartwright, 2002).
  Other Names: Xeloda

SUMMARY:
This study is a Phase 1b/2, dose-escalation, randomized, multicenter study to assess the efficacy, safety, tolerability, and PK of ivaltinostat in combination with capecitabine and capecitabine monotherapy in patients with metastatic pancreatic adenocarcinoma whose disease has not progressed on a first line fluoropyrimidine-based chemotherapy (e.g., FOLFIRINOX).

In Phase 1b, 3 dose levels of ivaltinostat will be studied in combination with a fixed dose of capecitabine to determine the RP2D of ivaltinostat.

In Phase 2, patients will be randomized in a 1:1 ratio to the combination of ivaltinostat and capecitabine or to capecitabine monotherapy. A fixed dose for capecitabine 1000 mg/m2 orally twice daily will be taken on Days 1 to 14, and the RP2D of ivaltinostat will be administered intravenously once a week for 2 weeks, followed by 1 week of rest. One cycle consists of 21 days. Tumor response during study treatment will be assessed every 6 weeks up to Cycle 10, then every 9 weeks afterwards using RECIST v1.1 criteria.

DETAILED DESCRIPTION:
There will be approximately 70 (18 Phase 1b dose-escalation, 52 Phase 2 randomized) patients in the study. In Phase 1b, 3 dose levels of ivaltinostat will be studied in combination with a fixed dose of capecitabine to determine the RP2D of ivaltinostat. In Phase 2, patients will be randomized in a 1:1 ratio to the combination of ivaltinostat and capecitabine or to capecitabine monotherapy as specified below:

Arm A

* Ivaltinostat (the dose will be selected after reviewing the results of Phase 1b among 3 dose levels of 60, 125, or 250 mg/m2) intravenous infusion over 60 minutes (±10 minutes) once on Days 1 and 8 of a 21-day cycle
* Capecitabine 1000 mg/m2 orally twice daily on Days 1 to 14 of a 21-day cycle OR Arm B
* Capecitabine 1000 mg/m2 orally twice daily on Days 1 to 14 of a 21-day cycle Study Assessments In Phase 1b, patients will attend clinic visits in Cycle 1 on Days 1, 2, 3, 5, 8, and 15 for assessments, with treatment on Days 1 and 8. After Cycle 1, patients will attend clinic visits on a weekly schedule for treatment (Days 1 and 8) and assessments (Days 1, 8, and 15) during 21-day cycles for the remainder of time receiving study treatment. In Phase 2, patients will attend clinic visits on a weekly schedule for treatment (Days 1 and 8) and assessments (Days 1, 8, and 15) during 21-day cycles.

The Phase 1b will enroll up to 18 patients (6 patients each of 3 dose levels of ivaltinostat [60, 125, and 250 mg/m2] + 1000 mg/m2 capecitabine BID) to assess the combination of ivaltinostat and capecitabine for safety and tolerability as well as to determine the ivaltinostat RP2D, assess the PDy of ivaltinostat, and assess PK parameters of both ivaltinostat and capecitabine. Data from the Phase 1b will be used in safety analyses but not in efficacy analyses.

Tumor response during study treatment will be assessed using RECIST v1.1 criteria. Baseline and on-treatment tumor assessments will be performed using CT or MRI scans with contrast of the chest, abdomen, and pelvis, with other regions as clinically indicated for the assessment of disease. Baseline evaluation should be performed within the 28-day screening period prior to the start of study treatment, as close as possible to randomization. Follow-up assessment consistent with baseline radiologic evaluation (i.e., if CT scan was performed for baseline assessment, then CT scan should be done for the follow-up evaluation) should be performed approximately every 6 weeks (±1 week) until objective disease progression as defined by RECIST v1.1. In addition to the imaging listed above, any other sites with known disease, or at which new disease is suspected, should also be appropriately imaged. Safety evaluations will occur at each protocol-specified study visit.

Patients will continue to receive study treatment until objective radiographic disease progression per RECIST v1.1 as assessed by the Investigator or until unacceptable toxicity occurs.

Once patients have discontinued study treatment, subsequent treatment options will be at the discretion of the treating physician. It is anticipated (but not required) that patients may be retreated with their first line regimen. Patients will be contacted on an approximately every-8-week schedule and followed up for survival. Details of any further anti-cancer treatment will be collected until death, loss to follow up, or withdrawal of consent. In addition to contact every 8 weeks, patients will be contacted in the 7 days following a specified date (data cut-off date) to capture survival status at that point for each survival analysis. Any patient who discontinues study treatment for reasons other than objective radiographic progression should continue to undergo scheduled objective tumor assessments according to the study plan in order to assess objective radiographic progression of disease.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years
* For Phase 1b, histologically or cytologically confirmed pancreatic adenocarcinoma (locally advanced or metastatic) with at least 1 prior therapy in either the advanced or perioperative setting
* For Phase 1b, measurable disease and/or non-measurable disease per RECIST v1.1
* For Phase 2, histologically or cytologically confirmed pancreatic adenocarcinoma without evidence of disease progression while receiving initial chemotherapy for metastatic disease (e.g., must have had a demonstrated CR, PR, or SD following initial chemotherapy).
* For Phase 2, measurable disease and/or non-measurable or no evidence of disease assessed by baseline CT (or MRI where CT is contraindicated). RECIST v1.1 will be used to allow for assessment of disease progression due to new lesions in patients with no evidence of disease at baseline. Patients with no evidence of disease following FOLFIRINOX chemotherapy will be deemed to have radiographic disease progression if new lesions are detected.
* For Phase 2, treatment with FOLFIRINOX for metastatic pancreatic adenocarcinoma at full or modified doses, for a minimum of 16 weeks, and no evidence of progression based on the radiographic imaging.
* a. Randomization must occur within 6 weeks of the last dose of chemotherapy.
* b. Patients who have received at least 16 weeks of FOLFIRINOX combination regimen but had non-fluoropyrimidine chemotherapeutic agents discontinued prior to 16 weeks due to toxicity are eligible if they have no radiographic evidence of disease.
* For Phase 2, patients who received prior chemotherapy or prior chemoradiation for a prior cancer or as adjuvant/neoadjuvant treatment for pancreatic adenocarcinoma are eligible provided at least 12 months have elapsed between the last dose of treatment and initiation of the FOLFIRINOX chemotherapy for metastatic pancreatic adenocarcinoma.
* Prior radiation therapy is allowed, provided >14 days have elapsed since completion of radiation prior to randomization.
* Adequate organ function
* ECOG Performance Status 0-1 at the date of signing the informed consent.

Exclusion Criteria:

* For Phase 2, radiographic progression of tumor per RECIST 1.1 between start of first line FOLFIRINOX chemotherapy for metastatic pancreatic adenocarcinoma and randomization.
* Cytotoxic chemotherapy or non-hormonal targeted therapy within 28 days of Cycle 1 Day 1 is not permitted. Palliative radiotherapy must have been completed 14 or more days before Cycle 1 Day 1. The patient can receive a stable dose of bisphosphonates or RANKL directed therapy for bone metastases before and during the study as long as these were initiated at least 2 weeks prior to study treatment
* For Phase 2, not receiving FOLFIRINOX as initial therapy for metastatic PDAC. Patients who received FOLFIRINOX initially and who needed to discontinue irinotecan or oxaliplatin due to toxicity are eligible, provided they received at least 4 weeks (2 cycles) of FOLFIRINOX
* For Phase 2, more than 1 prior line of therapy for metastatic PDAC
* Exposure to an investigational agent within 30 days or 5 half-lives (whichever is longer) prior to randomization
* Any previous treatment with a HDAC inhibitor, including ivaltinostat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) in phase 1 | 15 months
  The percentage of subjects who experience a grade 3 or higher adverse event that qualifies as a DLT
Incidence of treatment emergent AEs in phase 1 | 15 months
  The number of subjects who experience an adverse event that was possibly related to study drug
Treatment emergent changes in clinical laboratory tests in phase 1 | 15 months
  The number of subjects who experience a change in laboratory parameters that was possibly related to study drug.
Progression-Free Survival (PFS) in Phase 2 | 15 months
  Investigator assessed PFS

SECONDARY OUTCOMES:
Cmax of ivaltinostat in Phase 1 and 2 | 19 months
  Cmax will be assessed through the maximum measured plasma concentration occurring at Tmax
AUC of ivaltinostat in Phase 1 and 2 | 19 months
  Area under the plasma concentration (AUC) versus time curve from time 0 to time of least measurable concentration
Half-life (T1/2) of ivaltinostat in Phase 1 and 2 | 19 months
  Elimination half life will be calculated
Objective response rate (ORR) in Phase 1 and 2 | 19 months
  ORR per RECIST v1.1 Overall survival (OS).
Incidence of treatment emergent AEs in Phase 2 | 19 months
  The number of subjects who experience an adverse event that was possibly related to study drug

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H. Ko, MD, Principal Investigator — University of California, San Francisco
Locations (16):
- United States (16):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Hoag Medical Group, Newport Beach, California
  - UCSF Medical Center, San Francisco, California
  - UCLA Hematology/Oncology, Gastrointestinal Oncology, Santa Monica, California
  - University Cancer and Blood Center, Athens, Georgia
  - Community Health Network, Indianapolis, Indiana
  - Norton Cancer Institute Audubon, Louisville, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Clinical Research Alliance, Westbury, New York
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia